CLINICAL TRIAL: NCT06505733
Title: Postnatal Companion Support The Effect of Education on Maternal Depression and Fatigue: A Randomised Controlled Trial
Brief Title: Postnatal Companion Support The Effect of Education on Maternal Depression and Fatigue
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Huriye Altınkaynak, Chief Researcher, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KaratayU-EBE-HA-01
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Postpartum; Fatigue; Depression; Social Support
Keywords: social support; Depression; Fatigue; Postpartum
MeSH Terms: conditions — Fatigue; Depression

STUDY DESIGN:
Intervention Model Description: group who received companion training, group who did not receive training
Who Masked: Participant, Outcomes Assessor
Masking Description: The statistician will be blinded in the study. The researcher will not be blinded because he/she is the implementer. However, the researcher will open the envelope created by the statistician just before the application and learn which group the mother is in. In order to prevent bias in the evaluation of the data, the groups will be coded as A and B, and the data will be analysed by an independent statistician. After the analysis and interpretation of the data is completed, the codes of the intervention and control groups will be revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- attendants in the postnatal period (Experimental): In the guide, the needs of the postpartum mother and baby, postpartum depression (definition, symptoms, risk factors, complications, care), the role and responsibilities of the companion in supporting the postpartum mother are included.
  Interventions: Behavioral: postnatal attendant training
- non-intervention group (No Intervention): the group will not be trained

INTERVENTIONS:
Behavioral: postnatal attendant training — Intervention Group: Training and counselling will be provided to the puerperant and companions before discharge in a quiet and stimulus-free environment using the "Companion Training Guide". Research data will be collected three times: pre-test data, after the training and on the tenth day.
  Other Names: pre-test data, post-training and tenth day
  Arms: attendants in the postnatal period

SUMMARY:
In this study, it is aimed to investigate the effect of the trainings included in the content of the practical guide for postpartum supporter training companions, which will be given to the companions of women in the postpartum period, on depression and fatigue on mothers. The research will be conducted in methodological and single blind randomised control design. The study will be conducted at Necmettin Erbakan University Faculty of Medicine Hospital. A total of 70 puerperants will be included in the study as intervention (n: 35) and control (n: 35) groups. Introductory Information Form, Postpartum depression rating scale as data collection tools in the study: Motherhood Monitoring Scale by Parents (MMSP), Edinburgh Postnatal Depression Scale (EDDS), Multidimensional Fatigue Rating Scale will be used. The research data will be collected three times as pre-test data, fourth day and tenth day. Number, percentage, mean and standard deviation will be used in the evaluation of descriptive data; Chi-square test will be used for the similarity of the descriptive characteristics of the experimental and control groups; Kolmogrow-Smirnov and Shapiro-Wilk will be used in the normality analysis of dependent variables; t test in independent groups (student t test) will be used to compare the post-test scores of the experimental and control groups; and ANOVA in dependent groups will be used to compare the pre-test-post-test mean scores of the experimental group and eta square will be used to calculate effect sizes. The results obtained will be tested at p<0.05 significance level and bidirectionally. When the literature is examined, there is not enough data on the depression and fatigue of the companion caring for the woman in the postpartum period. This study aims to fill the gaps in the literature and to reduce depression and fatigue in mothers.

DETAILED DESCRIPTION:
One of the most important turning points in a woman's life is the pregnancy and birth process. In some cases, these milestones can turn into a crisis and lead to mental problems. In addition, for parents, preparing for and caring for a new baby is inherently a period of change and transition. With the addition of the responsibility of caring for the baby, more negative health problems may occur in the postpartum period. It is a risky period in terms of fatigue, emotional disorders, and postpartum depression during the transition to motherhood in the postpartum period. In the first three postnatal days, more than 50% of mothers experience maternal sadness, which is the mildest psychological disorder with symptoms of crying, sadness and unstable emotions. When this situation cannot be managed, postnatal depression occurs. According to previous research, 15% of mothers experience postnatal depression. The main symptoms of postnatal depression include lack of interest, low self-confidence, fatigue, sadness, sleep disturbance, loss of appetite, hostile attitude towards babies, self-blame and feelings of humiliation, and symptoms last for at least two weeks. Postnatal fatigue (PFF) is generally known to cause both a decrease in energy that prevents mothers from engaging in physical and mental activities after birth and impaired concentration and distraction that cannot be easily eliminated by rest or sleep. Edinburgh Postnatal Depression Scale is the gold standard for screening. The Turkish version has been used in Turkey since 1996 and the cut-off score is accepted as 13. In Turkey, the sensitivity of the scale is estimated to be 0.84 with a specificity of 0.88, indicating that 16% of women are overlooked for postnatal depression. It should be underlined that the scale is not routinely used in postnatal care and follow-up. In addition, it is difficult for women to diagnose themselves in terms of postnatal depression. Moreover, many mothers believe that they should not complain about the mental difficulties brought by the postnatal period. Therefore, self-assessment as well as the assessment of others is important.

In developed countries, almost all women and their babies receive labour and postnatal care. However, the quality and frequency of this care vary significantly. In developing countries, the need for care and support after birth remains unmet. Despite all its importance, this period is often the most neglected period. In the study conducted to evaluate the postnatal care services provided in family medicine units in terms of quantity and quality in our country, it is stated that although it is seen that postnatal care is provided at the level of developed countries in terms of quantity, the services provided in terms of content are insufficient, and the services provided should be evaluated not only in terms of quantity but also in terms of quality. PPF should provide physical relaxation by deliberately preventing and alleviating fatigue in the postpartum period with effective approaches. Postnatal care is defined as the most neglected aspect of maternity services and it is generally stated that less resources are allocated to it than antenatal care or delivery. Many developing countries with limited resources have difficulty in developing and implementing policies to prevent the treatment gap from increasing. Prevention or early detection and intervention programmes have been developed to reduce the burden of these two disorders. Effective community-based programmes have been shown to reduce depression. However, due to the lack of home visits in postnatal care services and inadequate quality, companion support is important in the postnatal period. Especially considering the quality of postnatal care in our country and the lack of home visits, the importance of companion support in this period comes to the fore. In a study examining the effect of companion support on acute stress reactions and postnatal depressive symptoms in the first three weeks after birth, it was reported that companion support reduced acute stress reactions and postnatal depressive symptoms. In a study, it is stated that companion support has a positive effect on the mother's mood and self-efficacy. In another study, it was stated that early and appropriate interventions to reduce PPF may increase the mitigation of negative effects on physical activity and therefore improve postnatal maternal health. In this period, the importance of the evaluation of the woman's own condition as well as the evaluation of health professionals and companions is emphasised. It is stated that observation of postnatal women by a close third person, especially by spouses and parents, will be beneficial.

Postnatal depression and fatigue are common problems in our country. However, postnatal care services are inadequate and unqualified. For this reason, studies should be carried out on alternative supports in postnatal care. In this context, "Postpartum Depression Parent Rating Scale for Postpartum Depression" was developed to increase the quality of early postnatal diagnosis and care: The Turkish validity and reliability study of the "Postpartum Depression Parent Rating Scale: Mother Monitoring Scale by Parents" and proving the effect of companion training on postpartum depression and fatigue constitute the original value of the project and our main motivation. The project has a unique value for a sustainable future in terms of its effects on the social level in terms of positive postnatal period and qualified support for puerperas and babies in general. In the project, ensuring that puerperas receive evidence and science-based postnatal support and care in line with our culture and traditions is also of unique value. It will also provide data for the comparison of innovative care models with traditional methods. Thus, it will help to improve, organise or develop capacity for future initiatives.

ELIGIBILITY:
Inclusion Criteria:

* Knowing how to read and write Turkish,
* Volunteer to participate in the research,
* She gave birth by cesarean section,
* Primiparous,
* Pregnant women who are open to communication (able to understand and answer questions) will be included in the sample.

Exclusion Criteria:

* Those who do not have the skills of reading, listening, writing, speaking and understanding Turkish,
* Those who have a hearing or visual impairment,
* Having postpartum complications,
* giving birth to stillbirth,
* People who wanted to withdraw from the study were not included.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — mother or mother-in-law of women in the postnatal period
Enrollment: 72 (Estimated)
Dates: Start 2024-08-07 (Estimated); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-08-17 (Estimated)

PRIMARY OUTCOMES:
change in the depression level of the companion on the 10th day of the postnatal period compared to the baseline value | 0-10 day
  The EPDS is a self-report scale consisting of 10 items in a 4-point Likert format. The responses consisting of four options are scored between 0-3, the lowest score that can be obtained from the scale is 0 and the highest score is 30. As the score increases, the level of depression increases. " Parent Rating Scale for Postpartum Depression: Maternity Monitoring Scale by Parents" , approval was received from the author after the translation of the scale questions.

SECONDARY OUTCOMES:
change in the fatigue level of the attendant on the 10th day of the postnatal period compared to the baseline value | 0-10 day
  ÇBYDS is a four-point Likert type scale consisting of 16 questions. As the score increases, his fatigue increases.

CONTACTS AND LOCATIONS:
Overall Officials: Hediye Ass. Prof. Karakoç, assistant professor, Study Director — KTO Karatay Univeristy

IPD SHARING:
Plan to Share IPD: Yes
yes
Supporting Information: Study Protocol
Time Frame: 7 August 2024-25 May 2025